CLINICAL TRIAL: NCT02237807
Title: Comparative, Randomized, Three -Period, Two-treatment, Three -Sequence, Open Label, Semi-replicate Crossover Bioequivalence Study of Dirithromycin 500 mg Enteric Coated Tablet (One Tablet) of (Abdi İbrahim İlaç San. Ve Tic. A. Ş., Turkey) Versus Dynabac 250 mg Enteric Coated Tablet (Two Tablets) of (Abdi İbrahim İlaç San. Ve Tic. A. Ş., Turkey) in Healthy Subjects Under Fed Conditions
Brief Title: Semi-replicate Crossover Bioequivalence Study of Dirithromycin in Healthy Subjects Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmaceutical Research Unit, Jordan (Other)
Collaborators: Abdi Ibrahim Ilac San. ve Tic A.S. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DIRI521/PRO-00
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Healthy
Keywords: Fed Conditions
MeSH Terms: interventions — dirithromycin; Tablets, Enteric-Coated

ARMS (2):
- DIRITHROMYCIN 500 MG ENTERIC COATED TABLET (Experimental): DIRITHROMYCIN 500 MG ENTERIC COATED TABLET of Abdi İbrahim İlaç San. Ve Tic. A. Ş., Turkey one tablet, once
  Interventions: Drug: DIRITHROMYCIN 500 MG ENTERIC COATED TABLET
- DYNABAC 250 MG ENTERIC COATED TABLET (Experimental): DYNABAC 250 MG ENTERIC COATED TABLET of Abdi İbrahim İlaç San. Ve Tic. A. Ş., Turkey, two tablets, once
  Interventions: Drug: DYNABAC 250 MG ENTERIC COATED TABLET

INTERVENTIONS:
Drug: DIRITHROMYCIN 500 MG ENTERIC COATED TABLET
  Arms: DIRITHROMYCIN 500 MG ENTERIC COATED TABLET
Drug: DYNABAC 250 MG ENTERIC COATED TABLET
  Arms: DYNABAC 250 MG ENTERIC COATED TABLET

SUMMARY:
The purpose of this study is to assess the bioequivalence of the investigational TEST product with the marketed REFERENCE products by measurement of Plasma concentrations of Erythromycylamine in plasma and calculation of the bioequivalence parameters from those measurements followed by ANOVA and 90% confidence interval statistical evaluation.

DETAILED DESCRIPTION:
An open-label, randomized, two-treatments, three-periods, three-sequences, semi-replicate crossover bioequivalence study with a washout period of at least 14 days between doses. Healthy, mixed skin Arab & Mediterranean Subjects ages between 18 and 50 years, body-mass index 18.5 to 30.0 kg/m2 inclusive (minimum of 50 kg weight), non-smokers or light smokers (smokers of not more than 10 cigarettes per day).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects.
2. Ethnic Group: Arab & Mediterranean.
3. Race: Mixed skin (white & black skin people).
4. Age 18-50 years.
5. Body-mass index 18.5 to 30.0 kg/m2 inclusive. (minimum of 50 kg weight)
6. Subject is available for the whole study period and gave written informed consent.
7. Normal Physical examination.
8. Vital signs within normal ranges.
9. All laboratory screening results within the normal range, or being assessed as clinically Non-significant by the attending physician.
10. Normal Kidney & Liver functions test

Exclusion Criteria:

1. Women of childbearing potential who don't use any contraceptive method, pregnant and/or lactating women.
2. Ethnic Group (Non- Arab &/ or Non- Mediterranean)
3. History of severe allergy or allergic reactions to study drug or related drugs or heparin
4. Known history or presence of food allergies, or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
5. History of serious illness that can impact fate of drugs
6. Known history or presence of cardiac, pulmonary, gastrointestinal, endocrine, musculoskeletal, neurological, hematological, liver or kidney disease.
7. Clinically significant illness 4 weeks before study Period I
8. Mental disease.
9. Smoking of more than 10 cigarettes per day
10. The intake of alcohol and grapefruit during the study.
11. The intake of caffeine, xanthenes, or CO2-containing beverages during hospitalization.
12. Regular use of medication.
13. Having taken medication that could affect the investigated drug product: a) Regular consumption of drugs during the two weeks prior to study initiation day, b) consumption of enzyme stimulating or inhibiting drugs (e.g. Barbiturates, Carbamazepine, Phenytoin, Amphetamine, Benzodiazepine, cannabinoid, cocaine, opiates, phencyclidine and methadone) during one month before the study initiation.
14. Presence of any significant physical or organ abnormality
15. Donation of 1) at least 400 ml of blood within 60 days, or 2) more than 150 ml of blood within 30 days, or 3) more than 100 ml blood plasma or platelets within 14 days before study Period I
16. Participation in another bioequivalence study and/or Clinical trials within 80 days prior to the start of this study Period I
17. Following a special diet (e.g. vegetarian) or dieting one month before the study initiation.
18. Subjects with seizures or prior history of seizures.
19. Prior history of hypersensitivity to dirithromycin, erythromycin, or other macrolide antibiotics
20. Any significant clinical abnormality including HBsAg, HCV, and / or HIV.
21. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration
22. Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
23. Exhausting physical exercise in the last 48 hours (e.g. weight lifting) or any recent significant change in dietary or exercise habits.
24. Subjects with history of Liver disease.
25. Abnormal Vital Signs.
26. Abnormal Kidney and/or Liver functions test.
27. Vomiting, Diarrhea on admission

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Cmax Ratio | pre-dosing and at 1.00, 2.00, 3.00, 3.50, 4.00, 4.50, 5.00, 5.50, 6.00, 6.50, 7.00, 8.00, 9.00, 10.00, 12.00, 14.00, 16.00, 20.00, 24.00, 36.00, 48.00, 72.00, 96.00 and 120.00 hours after dosing.
  Scaled average bioequivalence will be performed. Bioequivalence limits will be defined and widened according to the reference variance of σw2 within subject variability for the reference for Erythromycylamine.
AUC Ratio | pre-dosing and at 1.00, 2.00, 3.00, 3.50, 4.00, 4.50, 5.00, 5.50, 6.00, 6.50, 7.00, 8.00, 9.00, 10.00, 12.00, 14.00, 16.00, 20.00, 24.00, 36.00, 48.00, 72.00, 96.00 and 120.00 hours after dosing
  The 90% confidence interval for this measure lies within an acceptance range of 80.00% - 125.00%based on Erythromycylamine

CONTACTS AND LOCATIONS:
Overall Officials: Rana T Bustami, Phd.pharmacy, Principal Investigator — PRU
Locations (1):
- Arab Pharmaceutical industry Consulting/ Pharmaceutical Research Unit, Amman, Jordan